CLINICAL TRIAL: NCT03377790
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Pivotal Study to Evaluate the Safety and Efficacy of VP-102 Topical Film-Forming Solution [0.7% (w/v) Cantharidin] in Subjects (2 Years and Older) With Molluscum Contagiosum
Brief Title: Cantharidin Application in Molluscum Patients-1
Acronym: CAMP-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Verrica Pharmaceuticals Inc. (Industry)
Collaborators: Instat Consulting, Inc. (Other); Paidion Research, Inc. (Industry); Database Integrations, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-102-101
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Molluscum Contagiosum
Keywords: Molluscum; Skin Diseases; Poxviridae Infections; Skin Diseases; Infectious; Skin Diseases; Viral; DNA Poxvirus
MeSH Terms: conditions — Molluscum Contagiosum; Skin Diseases; Poxviridae Infections; Cellulitis; Skin Diseases, Viral | interventions — VP-102

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- VP-102 (Active Comparator): VP-102 is contained within a single-use applicator. The VP-102 applicator consists of a plastic tube containing a sealed glass ampule and an applicator tip. One ampule contains 450 μL of VP-102 (0.7% [w/v] cantharidin) solution.
  Interventions: Combination Product: VP-102 - Cantharidin, Topical Film Forming Solution
- Placebo (Placebo Comparator): Placebo is contained within a single-use applicator. The placebo applicator consists of a plastic tube containing a sealed glass ampule and an applicator tip. One ampule contains 450μl of placebo solution with the same color and consistency as VP-102.
  Interventions: Combination Product: Placebo -Topical Film Forming Solution without VP-102

INTERVENTIONS:
Combination Product: VP-102 - Cantharidin, Topical Film Forming Solution — VP-102, a single-use drug device combination product containing (cantharidin) topical solution, 0.7% (w/v). Up to 4 applications of VP-102 will be administered to Molluscum lesions at 21-day intervals.
  Arms: VP-102
Combination Product: Placebo -Topical Film Forming Solution without VP-102 — Placebo a single-use drug device combination product containing only the vehicle. Up to 4 applications of Placebo will be administered to Molluscum lesions at 21-day intervals.
  Arms: Placebo

SUMMARY:
This study is a Phase 3, randomized, double-blind, placebo-controlled, pivotal study to evaluate the safety and efficacy of VP-102 topical film-forming solution in subjects with Molluscum Contagiosum. VP-102 will be applied once every 21 days for up to 4 applications, to treatable molluscum contagiosum (molluscum) lesions on subjects 2 years and older. Efficacy will be assessed as the proportion of subjects achieving complete clearance of all treatable molluscum lesions (baseline and new) on the Day 84 visit.

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, randomized, double-blind, placebo (vehicle)-controlled, pivotal study that will be conducted in the United States to determine the efficacy and safety of VP-102 following treatment of molluscum lesions for up to 4 treatments, every 21 days, with VP-102/placebo in 250 subjects. Subjects will receive active VP-102 or placebo in a 3:2 ratio. Study drug (VP-102 or placebo) will be supplied in single-use applicators.

The film-forming Study drug solution will be applied and left on the lesions for 24 hours before the subject and/or parents/guardian washes the lesions. Study drug may be removed prior to the 24-hour time point in the event treatment-emergent AEs are experienced.

Molluscum lesions will be treated without occlusion in all anatomic areas including the face, trunk, back, arms, legs, hands, feet, anogenital region and buttocks.

ELIGIBILITY:
Inclusion Criteria:

To qualify for inclusion in this study, subjects must:

1. Be healthy subjects, at least 2 years of age or older.
2. Consent to having all molluscum lesions treated and the physician must be willing to treat all molluscum lesions initially present. Lesions within 10mm of the eyelid margins or the margin of any mucosal membrane should be evaluated carefully to ensure that they can be safely treated. Non-mucosal genital area lesions and inflamed lesions are considered treatable.
3. Be otherwise medically healthy with no clinically significant medical history as determined by the investigator. Subjects exhibiting active Atopic Dermatitis may be enrolled.
4. On day of treatment refrain from application of all topical agents including alcohol-based sanitary products and sunscreens for a minimum of 4 hours before Study drug application. Topical agents including alcohol-based sanitary products and sunscreens may be used after application of the study drug so long as they are not applied within 5cm of treated skin lesions.
5. Refrain from swimming, bathing or prolonged immersion in water or any liquids until the Study drug is removed.
6. Have the ability or have a guardian with the ability to follow study instructions and be likely to complete all study requirements.
7. Provide written informed consent or assent in a manner approved by the institutional review board (IRB) and/or have a parent/guardian provide written informed consent as evidenced by the signature on an IRB approved assent/consent form.
8. Provide written authorization for use and disclosure of protected health information.
9. Agree to allow photographs to be taken, (selected sites only) of selected lesions at every visit that will be used for training, publication and future marketing brochures.

Exclusion Criteria:

Subjects will be excluded from the study if they:

1. Are unable to cooperate with the requirements or visits of the study, as determined by the investigator.
2. Are systemically immunosuppressed or are receiving treatments such as chemotherapy or other non-topical immunosuppressive agents.
3. Have any lesions present at baseline in anatomic locations that the subject/parent/guardian or the physician is unwilling to treat.
4. Have had any previous treatment of molluscum including the use of cantharidin, antivirals, retinoids, curettage or freezing of lesions in the past 14 days. Additional treatments should not be implemented during the course of the study.
5. Have a history of illness or any dermatologic disorder which, in the opinion of the investigator, will interfere with accurate counting of lesions or increase the risk of adverse events.
6. History or presence of clinically significant medical, psychiatric, or emotional condition or abnormality that, in the opinion of the investigator, would compromise the safety of the subject or the quality of the data.
7. Have a history or presence of hypersensitivity or an idiosyncratic reaction to the Study drug or related compounds, or drug product excipients (acetone, ethyl alcohol, nitrocellulose, hydroxypropyl cellulose, castor oil, camphor, gentian violet, and denatonium benzoate).
8. Have a condition or situation that may interfere significantly with the subject's participation in the study (e.g., subjects who required hospitalization in the 2 months prior to screening for an acute or chronic condition including alcohol or drug abuse), at the discretion of the investigator.
9. Have received another investigational product within 14 days prior to the first application of the Study drug.
10. Have been treated within 14 days with a product that contains cantharidin (topical or homeopathic preparations) for any reason prior to screening.
11. Are sexually active or may become sexually active and are unwilling to practice responsible birth control methods. (e.g., combination of condoms and foam, birth control pills, intrauterine device, patch, shot and vaginal ring, etc.). Withdrawal is not an acceptable method of birth control. Females that have reached menarche must have a negative urine pregnancy test at each visit prior to treatment with Study drug.
12. Are pregnant or breastfeeding.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Eichenfield, MD, Principal Investigator — Rady Children's Hospital; San Diego, California
Locations (18):
- United States (18):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Southeastern Pediatric Associates, Dothan, Alabama
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Study Protocol, Inc.,, Boynton Beach, Florida
  - Skin Research Institute, Coral Gables, Florida
  - ASCLEPES Research Center, Spring Hill, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Summit Dermatology, Oakbrook Terrace, Illinois
  - Clarkston Skin Research, Clarkston, Michigan
  - St Louis Children's Hospital, St Louis, Missouri
  - Midwest Children's Hospital, Lincoln, Nebraska
  - Kings County Hospital, Brooklyn, New York
  - University North Carolina Dermatology Center, Chapel Hill, North Carolina
  - The Pediatric Associates of Fairfield, Inc, Fairfield, Ohio
  - Holston Medical Group, Bristol, Tennessee
  - Arlington Research Center, Arlington, Texas
  - Center for Skin Research, Houston, Texas
  - ACRC Trials Plano Pediatrics, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eichenfield LF, Kwong P, Gonzalez ME, Yan A, D'Arnaud P, Burnett P, Olivadoti M. Safety and Efficacy of VP-102 (Cantharidin, 0.7% w/v) in Molluscum Contagiosum by Body Region: Post hoc Pooled Analyses from Two Phase III Randomized Trials. J Clin Aesthet Dermatol. 2021 Oct;14(10):42-47. PMID 34976290
- [Derived] Eichenfield LF, Siegfried E, Kwong P, McBride M, Rieger J, Glover D, Willson C, Davidson M, Burnett P, Olivadoti M. Pooled Results of Two Randomized Phase III Trials Evaluating VP-102, a Drug-Device Combination Product Containing Cantharidin 0.7% (w/v) for the Treatment of Molluscum Contagiosum. Am J Clin Dermatol. 2021 Mar;22(2):257-265. doi: 10.1007/s40257-020-00570-8. Epub 2021 Feb 18. PMID 33599960
- [Derived] Eichenfield LF, McFalda W, Brabec B, Siegfried E, Kwong P, McBride M, Rieger J, Willson C, Davidson M, Burnett P. Safety and Efficacy of VP-102, a Proprietary, Drug-Device Combination Product Containing Cantharidin, 0.7% (w/v), in Children and Adults With Molluscum Contagiosum: Two Phase 3 Randomized Clinical Trials. JAMA Dermatol. 2020 Dec 1;156(12):1315-1323. doi: 10.1001/jamadermatol.2020.3238. PMID 32965495

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pre-study screening for eligibility (ICF and assent, [when applicable], demographics, physical exam, prior and concomitant meds and molluscum and medical hx) could occur up to 14 days before, or on the same day as Study drug application. Subjects not meeting criteria at Treatment Visit 1 were to be discontinued and treated per standard of care. Note: 2 subjects randomized to placebo received VP-102 were included in VP-102 for Safety. There was one subject randomized to VP-102 but not treated.
Groups:
- VP-102: VP-102 Film Forming Solution applied via a prefilled applicator to affected area every 21 days
  VP-102: VP-102, a single-use drug device combination product containing (cantharidin) topical solution, 0.7% (w/v). VP-102 Active will be administered to Molluscum lesions
- Placebo: Vehicle Film Forming Solution applied via a prefilled applicator to affected area every 21 days
  Placebo: Placebo a single-use drug device combination product containing only the vehicle will be administered to Molluscum lesions
Period: Overall Study
Arm/Group | VP-102 | Placebo
Started | 160 | 106
Completed | 150 | 100
Not Completed | 10 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Randomized but not treated | 1 | 0
Not completed — Withdrawn by Parent/Guardian | 7 | 4

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | VP-102 | Placebo | Total
Number analyzed (Participants) | 160 | 106 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.5 (5.29) | 6.3 (4.67) | 7.4 (5.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 61 | 146
  Male | 75 | 45 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 8 | 28
  Not Hispanic or Latino | 140 | 98 | 238
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 5 | 15
  White | 135 | 98 | 233
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 2 | 13
Region of Enrollment [Number; unit: participants]
  United States | 160 | 106 | 266
Baseline number of treatable molluscum lesions [Mean (Standard Deviation); unit: molluscum lesions] | 22.2 (23.12) | 24.8 (24.97) | 23.2 (23.86)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Exhibiting Complete Clearance of All Treatable Molluscum Lesions (Baseline and New) on the Day 84 Visit (EOS)
Description: Percentage of subjects exhibiting complete clearance of all treatable molluscum lesions (baseline and new) on the Day 84 visit (EOS).
Time Frame: Day 1 (Baseline and new) compared to Day 84 (EOS)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | VP-102 | Placebo
Number analyzed (Participants) | 160 | 106
Participants | 74 | 19
Statistical Analysis 1: Comparison: VP-102 vs Placebo; Test type: Superiority; p < 0.0001, Chi-squared — Differences between treatments arms are compared using a chi-square test

2. Secondary Outcome: Percentage of Subjects Exhibiting Complete Clearance of All Treatable Molluscum Lesions (Baseline and New) on the Day 63 Visit
Description: Percentage of subjects exhibiting complete clearance of all treatable molluscum lesions (baseline and new) on the Day 63 visit.
Time Frame: Day 1 (Baseline and new) compared to Day 63
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | VP-102 | Placebo
Number analyzed (Participants) | 160 | 106
Participants | 51 | 18
Statistical Analysis 1: Comparison: VP-102 vs Placebo; Test type: Superiority; p = 0.0067, Chi-squared; Differences between treatments arms are compared using a chi-square test

3. Secondary Outcome: Percentage of Subjects Exhibiting Complete Clearance of All Treatable Molluscum Lesions (Baseline and New) on the Day 42 Visit
Description: Percentage of subjects exhibiting complete clearance of all treatable molluscum lesions (baseline and new) on the Day 42 visit.
Time Frame: Day 1 (Baseline and new) compared to Day 42
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | VP-102 | Placebo
Number analyzed (Participants) | 160 | 106
Participants | 33 | 10
Statistical Analysis 1: Comparison: VP-102 vs Placebo; Test type: Superiority; p = 0.0152, Chi-squared; Differences between treatments arms are compared using a chi-square test

4. Secondary Outcome: Proportion of Subjects Exhibiting Complete Clearance of All Treatable Molluscum Lesions (Baseline and New) on the Day 21 Visit
Description: Proportion of subjects exhibiting complete clearance of all treatable molluscum lesions (baseline and new) on the Day 21 visit.
Time Frame: Day 1 (Baseline and new) compared to Day 21
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | VP-102 | Placebo
Number analyzed (Participants) | 160 | 106
Participants | 18 | 4
Statistical Analysis 1: Comparison: VP-102 vs Placebo; Test type: Superiority; p = 0.0302, Chi-squared; Differences between treatments arms are compared using a chi-square test

5. Other Pre Specified Outcome: Change From Baseline to EOS Day 84 of the Composite Score From the Children's Dermatology Life Quality Index (CDLQI) Assessment at the EOS Visit to Measure the Quality of Life and Impact of Skin Disease in the Subset of Subjects 4 -16 Years of Age.
Description: Change from Baseline to EOS Day 84 of the Composite Score From the Children's Dermatology Life Quality Index (CDLQI) Assessment at the EOS Visit to Measure the Quality of Life and Impact of Skin Disease in the Subset of Subjects 4 -16 Years of Age.
  From responses to that questionnaire, a composite score was calculated. The calculated composite score was the sum of the individual 10 items of the CDLQI and could range from 0-30. For each item on the
  CDLQI, a score of 0-3 was assigned using the following scores per response:
  * 3: Very much (or Prevented School, Question 7 only)
  * 2: Quite a lot
  * 1: Only a little
  * 0: Not at all Larger composite CDLQI scores indicate skin condition is having more effect on subjects' lives (worse outcome).
Time Frame: Baseline to Day 84 (EOS)
Population: ITT Population (Subjects 4-16 years of age)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VP-102 | Placebo
Number analyzed (Participants) | 122 | 78
units on a scale | -2.1 (2.70) | -2.7 (3.46)
Statistical Analysis 1: Comparison: VP-102 vs Placebo; Test type: Superiority; p = 0.5921, ANCOVA; Differences between Tx arms are compared using an ANCOVA with treatment as the independent factor and baseline CDLQI composite score as the covariate

6. Other Pre Specified Outcome: Percent Change of All Treatable Molluscum Lesions (Baseline and New) From Baseline at the EOS Visit
Description: Percent change of all treatable molluscum lesions (baseline and new) from baseline at the EOS visit.
Time Frame: Day 1 (Baseline) compared to Day 84 (EOS)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percentage of change in wart count
Arm/Group | VP-102 | Placebo
Number analyzed (Participants) | 157 | 104
percentage of change in wart count | -69.2 (98.13) | 20.0 (239.72)
Statistical Analysis 1: Comparison: VP-102 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Differences between treatment arms are compared using an ANCOVA, with treatment as the independent factor and baseline lesion count as the covariate

7. Other Pre Specified Outcome: Change From Baseline in the Number of Treatable Molluscum Lesions (Baseline and New) at the EOS Visit.
Description: Change from baseline in the number of treatable molluscum lesions (baseline and new) at the EOS visit.
Time Frame: Day 1 (Baseline) compared to Day 84 (EOS)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: change in wart count
Arm/Group | VP-102 | Placebo
Number analyzed (Participants) | 157 | 104
change in wart count | -18.3 (22.64) | -5.9 (33.33)
Statistical Analysis 1: Comparison: VP-102 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 6, analysis 1]

8. Other Pre Specified Outcome: Percentage of Subjects Exhibiting a 75% or Greater Reduction of All Treatable Molluscum Lesions (Baseline and New) at the EOS Visit.
Description: Percentage of subjects that exhibited a 75% or greater clearance of all treatable molluscum lesions (baseline and new) at the EOS visit.
Time Frame: Day 1 (Baseline) compared to Day 84 (EOS)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | VP-102 | Placebo
Number analyzed (Participants) | 160 | 106
Participants | 119 | 36
Statistical Analysis 1: Comparison: VP-102 vs Placebo; Test type: Superiority; p < 0.0001, Chi-squared; Differences between treatments arms are compared using a chi-square test

9. Other Pre Specified Outcome: Percentage of Subjects Exhibiting a 90% or Greater Reduction of All Treatable Molluscum Lesions (Baseline and New) at the EOS Visit.
Description: Percentage of subjects that exhibited a 90% or greater clearance of all treatable molluscum lesions (baseline and new) at the EOS visit.
Time Frame: Day 1 (Baseline) compared to Day 84 (EOS)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | VP-102 | Placebo
Number analyzed (Participants) | 160 | 106
Participants | 99 | 28
Statistical Analysis 1: Comparison: VP-102 vs Placebo; Test type: Superiority; p < 0.0001, Chi-squared; Differences between treatments arms are compared using a chi-square test

10. Other Pre Specified Outcome: Subject Reported Spread to Household Members as Measured by Any New Occurrence of Molluscum in Household Members of Subject.
Description: Subject reported spread to household members as measured by any new occurrence of molluscum in household members of subject. To be eligible for assessment, subjects had to have at least one household member free of lesions at baseline and have at least 1 post baseline assessment of spread of molluscum lesions.
Time Frame: Days 1, 21, 42, 63 and 84 (EOS).
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | VP-102 | Placebo
Number analyzed (Participants) | 160 | 106
Participants | 9 | 13
Statistical Analysis 1: Comparison: VP-102 vs Placebo; Test type: Superiority; p = 0.0520, Chi-squared; Differences between treatments arms are compared using a chi-square test

ADVERSE EVENTS:
Time Frame: Treatment Visit 1 up to 30 days after EOS Day Visit.
Description: Note: Related TEAE= TEAEs with relationship of Definitely, Probably or Possibly Related or have a missing relationship.
  Note: A Local Skin Reaction TEAE is defined as any Targeted AE that was identified as a Related AE.
  Note: 2 subjects randomized to placebo received VP-102 were included in VP-102 for Safety. There was one subject randomized to VP-102 but not treated.)
Arm/Group | VP-102 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/161 | 1/104
Other Adverse Events (participants affected / at risk) | 159/161 | 76/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VP-102 (N=161) | Placebo (N=104)
Serious Treatment Emergent Adverse Events (Surgical and medical procedures) | 0 (0) | 1 (1) — Appendicectomy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VP-102 (N=161) | Placebo (N=104)
Application site pruritus (Skin and subcutaneous tissue disorders) | 104 | 38
Application site erythema (Skin and subcutaneous tissue disorders) | 69 | 30
Application site scab (Skin and subcutaneous tissue disorders) | 62 | 25
Application site discolouration (Skin and subcutaneous tissue disorders) | 54 | 18
Application site dryness (Skin and subcutaneous tissue disorders) | 24 | 11
Application site erosion (Skin and subcutaneous tissue disorders) | 10 | 2
Application site scar (Skin and subcutaneous tissue disorders) | 7 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 5
Application site vesicles (Skin and subcutaneous tissue disorders) | 157 | 29
Application site pain (Injury, poisoning and procedural complications) | 110 | 20
Application site oedema (Injury, poisoning and procedural complications) | 21 | 6
Pharyngitis streptococcal (Infections and infestations) | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is bound to terms and conditions of a Sponsored Clinical Trial Agreement which has strict confidentiality obligations running to Sponsor and broad provisions restricting PI's rights to publish or present any data or Study Results without Sponsor's express review consent and review.

DOCUMENTS (2):
  • Study Protocol (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT03377790/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT03377790/SAP_001.pdf